CLINICAL TRIAL: NCT03681886
Title: Evaluation of Visual and Refractive Outcomes of The ClarVista HARMONI™ Modular Intraocular Lens System
Brief Title: Visual and Refractive Outcomes of The ClarVista HARMONI™ Modular Intraocular Lens System (HMIOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ClarVista Medical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CVM-00001
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Cataract; Aphakia
Keywords: intraocular lens; IOL; intraoperative exchange
MeSH Terms: conditions — Cataract; Aphakia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Primary Implantation (Cohort 1) (Experimental): Primary implantation with HMIOL through Month 1 visit, followed by study exit. 1 site followed up to Month 12.
  Interventions: Device: Harmoni Modular Intraocular Lens
- Optic Exchange (Cohort 2) (Experimental): Subset of Cohort 1 with optic exchange at Month 1 post primary implantation, followed up to Month 1 post optic exchange
  Interventions: Device: Harmoni Modular Intraocular Lens; Procedure: Optic Exchange

INTERVENTIONS:
Device: Harmoni Modular Intraocular Lens — Two-component system consisting of a base and a separate optic that allows for an intraoperative exchange of the optic only without direct manipulation of the capsular bag.
  Other Names: HMIOL
Procedure: Optic Exchange — Removal of one optic and replacement with another for the purpose of improving refractive outcomes
  Arms: Optic Exchange (Cohort 2)

SUMMARY:
The purpose of this study was to evaluate visual and refractive outcomes with the use of the HARMONI™ Modular Intraocular Lens (HMIOL) System implantation, assembly, and optic exchange in subjects undergoing cataract surgery.

DETAILED DESCRIPTION:
All subjects were implanted with the HARMONI™ Modular Intraocular Lens (HMIOL) System in the right eye, left eye, or both eyes based on the best interest of the subject and the clinical judgment the Investigator (Day 0, primary implantation) (Cohort 1). At Month 1 post primary implantation, subjects were given the option to undergo an optic exchange procedure. Subjects who underwent the optic exchange (Cohort 2) (Day 0, optic exchange) were followed for an additional month. Subjects who did not undergo an optic exchange were exited from the study, except at 1 site, which followed subjects up to Month 12.

Alcon Research, LLC, acquired ClarVista Medical in 2017. This study was designed and conducted by ClarVista Medical, Inc. The study results were collected, analyzed, and provided by ClarVista Medical, Inc. to Alcon Research, LLC.

ELIGIBILITY:
Key Inclusion Criteria:

* Able to understand and sign an approved Informed Consent Form (ICF);
* Willing and able to return for scheduled treatment and follow-up examinations;
* Planned removal of cataracts (cortical, nuclear, subcapsular, or a combination) by manual phacoemulsification cataract extraction;

Key Exclusion Criteria:

* Any ocular conditions which could affect the stability of the IOL in either eye;
* Traumatic or congenital cataract;
* Pregnancy or planned pregnancy during the study period;
* Medications that may confound the outcome or increase risk to the subject;
* Any clinical finding or intraocular complication during primary cataract surgery or Implantation of the lens system likely to increase complications or risk to the subject;
* Other protocol-specified exclusion criteria may apply.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-01-09 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Surgical, Study Director — Alcon Research, LLC

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 5 Investigators participated in the study; 3 in the Philippines, 1 in Mexico, and 1 in Panama.
Pre-assignment Details: Of the 150 subjects enrolled, 72 were exited from the study prior to attempted implantation with the HARMONI™ Modular Intraocular Lens (HMIOL) System. This reporting group includes all subjects / eyes with attempted implantation.
Units Other Than Participants: eyes
Groups:
- All HMIOL Cohort: Implantation of the HARMONI™ Modular Intraocular Lens (HMIOL) System in the right eye, left eye, or both eyes
Period: Overall Study
Arm/Group | All HMIOL Cohort
Started | 78; 100 eyes
Successful Implantation | 76; 98 eyes
Failed Implantation | 2; 2 eyes
Underwent Optic Exchange | 4; 4 eyes
Completed | 76; 98 eyes
Not Completed | 2; 2 eyes

BASELINE CHARACTERISTICS:
Population: Safety Population: All subjects/eyes with attempted HMIOL implantation (successful or aborted after contact with the eye)
Groups:
- All HMIOL Cohort: All subjects with attempted implantation of the HARMONI™ Modular Intraocular Lens (HMIOL) System in the right eye, left eye, or both eyes
Arm/Group | All HMIOL Cohort
Number analyzed (Participants) | 78
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.4 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 31
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 50
  Black | 0
  Caucasian | 0
  Other | 28

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eyes With Uncorrected Distance Visual Acuity (UCDVA) by Visit - Cohort 1
Description: Visual acuity of the eye was tested while reading charts at 20-foot equivalent distance from the participant with an optical infinity adjustment of +0.25 diopter (D). UCDVA was recorded in Snellen, with 20/20 considered to be 'normal' vision. A visual acuity of 20/40 means the participant is able to read a certain size letter 20 feet away that a person with 'normal' vision would be able to read from 40 feet away. A larger denominator, therefore, indicates a lower visual acuity. No formal statistical hypothesis testing was planned.
Time Frame: Day 1 post primary implantation, Week 1 post primary implantation, Month 1 post primary implantation, Month 3 post primary implantation, Month 6 post primary implantation, Month 12 post primary implantation
Population: Per Protocol: All subjects/eyes with successful implantation of HMIOL with no major protocol deviations and available data.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Cohort 1 - Day 1 Post Primary Implantation; Cohort 1 - Week 1 Post Primary Implantation; Cohort 1 - Month 1 Post Primary Implantation; Cohort 1 - Month 3 Post Primary Implantation; Cohort 1 - Month 6 Post Primary Implantation; Cohort 1 - Month 12 Post Primary Implantation: Primary implantation with HMIOL through Month 1 visit, followed by study exit. 1 site followed up to Month 12.
Arm/Group | Cohort 1 - Day 1 Post Primary Implantation | Cohort 1 - Week 1 Post Primary Implantation | Cohort 1 - Month 1 Post Primary Implantation | Cohort 1 - Month 3 Post Primary Implantation | Cohort 1 - Month 6 Post Primary Implantation | Cohort 1 - Month 12 Post Primary Implantation
Number analyzed (Participants) | 74 | 75 | 75 | 12 | 12 | 12
Number analyzed (eyes) | 96 | 97 | 97 | 12 | 12 | 12
percentage of eyes
  20/20 Snellen or Better | 30.2 | 32.0 | 32.0 | 16.7 | 58.3 | 25.0
  20/25 Snellen or Better | 53.1 | 61.9 | 60.8 | 58.3 | 83.3 | 50.0
  20/32 Snellen or Better | 74.0 | 84.5 | 78.4 | 91.7 | 91.7 | 66.7
  20/40 Snellen or Better | 85.4 | 89.7 | 93.8 | 91.7 | 100.0 | 100.0
  Worse than 20/40 Snellen | 14.6 | 10.3 | 6.2 | 3.3 | 0.0 | 0.0

2. Primary Outcome: Percentage of Eyes With Uncorrected Distance Visual Acuity (UCDVA) by Visit - Cohort 2
Description: Visual acuity of the eye was tested while reading charts at 20-foot equivalent distance from the participant with an optical infinity adjustment of +0.25 diopter (D). UCDVA was recorded in Snellen, with 20/20 considered to be 'normal' vision. A visual acuity of 20/40 means the participant is able to read a certain size letter 20 feet away that a person with 'normal' vision would be able to read from 40 feet away. A larger denominator, therefore, indicates a lower visual acuity. No formal statistical hypothesis testing was planned. The optic exchange occurred 1 month following primary implantation with HMIOL.
Time Frame: Day 0 pre optic exchange, Day 1 post optic exchange, Week 1 post optic exchange, Month 1 post optic exchange
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Cohort 2 - Day 0 Pre Optic Exchange; Cohort 2 - Day 1 Post Optic Exchange; Cohort 2 - Week 1 Post Optic Exchange; Cohort 2 - Month 1 Post Optic Exchange: Subset of Cohort 1 with optic exchange at Month 1 post primary implantation, followed up to Month 1 post optic exchange
Arm/Group | Cohort 2 - Day 0 Pre Optic Exchange | Cohort 2 - Day 1 Post Optic Exchange | Cohort 2 - Week 1 Post Optic Exchange | Cohort 2 - Month 1 Post Optic Exchange
Number analyzed (Participants) | 3 | 3 | 3 | 3
Number analyzed (eyes) | 3 | 3 | 3 | 3
percentage of eyes
  20/20 Snellen or Better | 0.0 | 66.7 | 66.7 | 66.7
  20/25 Snellen or Better | 0.0 | 66.7 | 66.7 | 66.7
  20/32 Snellen or Better | 0.0 | 66.7 | 100.0 | 100.0
  20/40 Snellen or Better | 66.7 | 100.0 | 100.0 | 100.0
  Worse than 20/40 Snellen | 33.3 | 0.0 | 0.0 | 0.0

3. Primary Outcome: Percentage of Eyes With Best Corrected Distance Visual Acuity (BCDVA) by Visit - Cohort 1
Description: Visual acuity of the eye was tested while reading charts at 20-foot equivalent distance from the participant with subject manifest refraction in place. BCDVA was recorded in Snellen, with 20/20 considered to be 'normal' vision. A visual acuity of 20/40 means the participant is able to read a certain size letter 20 feet away that a person with 'normal' vision would be able to read from 40 feet away. A larger denominator, therefore, indicates a lower visual acuity. No formal statistical hypothesis testing was planned.
Time Frame: Baseline (Day -90 to Day 0 preoperative), Week 1 post primary implantation, Month 1 post primary implantation, Month 3 post primary implantation, Month 6 post primary implantation, Month 12 post primary implantation
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Cohort 1 - Baseline (Day -90 to Day 0 Preoperative); Cohort 1 - Week 1 Post Primary Implantation; Cohort 1 - Month 1 Post Primary Implantation; Cohort 1 - Month 3 Post Primary Implantation; Cohort 1 - Month 6 Post Primary Implantation; Cohort 1 - Month 12 Post Primary Implantation: Primary implantation with HMIOL through Month 1 visit, followed by study exit. 1 site followed up to Month 12.
Arm/Group | Cohort 1 - Baseline (Day -90 to Day 0 Preoperative) | Cohort 1 - Week 1 Post Primary Implantation | Cohort 1 - Month 1 Post Primary Implantation | Cohort 1 - Month 3 Post Primary Implantation | Cohort 1 - Month 6 Post Primary Implantation | Cohort 1 - Month 12 Post Primary Implantation
Number analyzed (Participants) | 71 | 75 | 75 | 12 | 12 | 12
Number analyzed (eyes) | 92 | 97 | 97 | 12 | 12 | 12
percentage of eyes
  20/20 Snellen or Better | 13.0 | 76.3 | 72.2 | 83.3 | 91.7 | 58.3
  20/25 Snellen or Better | 23.9 | 83.5 | 92.8 | 100.0 | 100.0 | 91.7
  20/32 Snellen or Better | 44.6 | 94.8 | 96.9 | 100.0 | 100.0 | 100.0
  20/40 Snellen or Better | 58.7 | 96.9 | 99.0 | 100.0 | 100.0 | 100.0
  Worse than 20/40 Snellen | 41.3 | 3.1 | 1.0 | 0.0 | 0.0 | 0.0

4. Primary Outcome: Percentage of Eyes With Best Corrected Distance Visual Acuity (BCDVA) by Visit - Cohort 2
Description: as for outcome 3
Time Frame: Baseline (Day 0 pre optic exchange), Week 1 post optic exchange, Month 1 post optic exchange
Population: as for outcome 1
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Cohort 2 - Baseline (Day 0 Pre Optic Exchange),; Cohort 2 - Week 1 Post Optic Exchange; Cohort 2 - Month 1 Post Optic Exchange: Subset of Cohort 1 with optic exchange at Month 1 post primary implantation, followed up to Month 1 post optic exchange
Arm/Group | Cohort 2 - Baseline (Day 0 Pre Optic Exchange), | Cohort 2 - Week 1 Post Optic Exchange | Cohort 2 - Month 1 Post Optic Exchange
Number analyzed (Participants) | 3 | 3 | 3
Number analyzed (eyes) | 3 | 3 | 3
percentage of eyes
  20/20 Snellen or Better | 33.3 | 100.0 | 66.7
  20/25 Snellen or Better | 66.7 | 100.0 | 100.0
  20/32 Snellen or Better | 100.0 | 100.0 | 100.0
  20/40 Snellen or Better | 100.0 | 100.0 | 100.0
  Worse than 20/40 Snellen | 0.0 | 0.0 | 0.0

5. Primary Outcome: Mean Manifest Refraction Spherical Equivalent (MRSE) by Visit - Cohort 1
Description: A manifest refraction (manual vision test) was conducted using letter charts and a phoropter. The subject was manually refracted to his/her best correction. The manifest refraction spherical equivalent (MRSE) was measured in diopters (D) and calculated as follows: sphere + 1/2 cylinder. A less negative value indicates a more accurate IOL power calculation. No formal statistical hypothesis testing was planned.
Time Frame: as for outcome 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Arm/Group | Cohort 1 - Baseline (Day -90 to Day 0 Preoperative) | Cohort 1 - Week 1 Post Primary Implantation | Cohort 1 - Month 1 Post Primary Implantation | Cohort 1 - Month 3 Post Primary Implantation | Cohort 1 - Month 6 Post Primary Implantation | Cohort 1 - Month 12 Post Primary Implantation
Number analyzed (Participants) | 75 | 75 | 75 | 12 | 12 | 12
Number analyzed (eyes) | 97 | 97 | 97 | 12 | 12 | 12
diopter | -0.53 (2.70) | -0.28 (0.62) | -0.29 (0.63) | -0.58 (0.57) | -0.49 (0.61) | -0.40 (0.69)

6. Primary Outcome: Mean Manifest Refraction Spherical Equivalent (MRSE) by Visit - Cohort 2
Description: as for outcome 5
Time Frame: Baseline (Day 0 pre optic exchange), Week 1 post optic exchange, Month 1 post optic exchange
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: diopter
Units Other Than Participants: eyes
Groups:
- Cohort 2 - Baseline (Day 0 Pre Optic Exchange); Cohort 2 - Week 1 Post Optic Exchange; Cohort 2 - Month 1 Post Optic Exchange: Subset of Cohort 1 with optic exchange at Month 1 post primary implantation, followed up to Month 1 post optic exchange
Arm/Group | Cohort 2 - Baseline (Day 0 Pre Optic Exchange) | Cohort 2 - Week 1 Post Optic Exchange | Cohort 2 - Month 1 Post Optic Exchange
Number analyzed (Participants) | 3 | 3 | 3
Number analyzed (eyes) | 3 | 3 | 3
diopter | -1.54 (0.56) | -0.25 (0.25) | -0.17 (0.29)

7. Primary Outcome: Number of Surgeon Responses to Primary Surgery Question: How Would You Rate the Surgical Difficulty of the Base Implantation? - All HMIOL Cohort
Description: The surgeon's response was collected on a study-specific questionnaire after each surgery. No formal statistical hypothesis testing was planned.
Time Frame: Day 0 primary implantation
Population: Safety Population: All eyes with attempted HMIOL implantation (successful or aborted after contact with the eye) and available data
Measure: Number; unit: surgeon response
Units Other Than Participants: eyes
Groups:
- All HMIOL Cohort: Primary implantation with HMIOL
Arm/Group | All HMIOL Cohort
Number analyzed (Participants) | 76
Number analyzed (eyes) | 98
surgeon response
  Easier than a traditional single piece IOL | 35
  Slightly easier than a traditional single piece IO | 16
  The same as a traditional single piece IOL | 11
  Slightly more difficult than a trd'l single pc IOL | 34
  More difficult than a traditional single piece IOL | 2

8. Primary Outcome: Number of Surgeon Responses to Primary Surgery Question: How Would You Rate the Surgical Difficulty of the Optic Implantation and Assembly? - All HMIOL Cohort
Description: as for outcome 7
Time Frame: Day 0 primary implantation
Population: as for outcome 7
Measure: Number; unit: surgeon response
Units Other Than Participants: eyes
Arm/Group | All HMIOL Cohort
Number analyzed (Participants) | 76
Number analyzed (eyes) | 98
surgeon response
  Very easy | 31
  Easy | 23
  Neutral | 35
  Difficult | 8
  Very difficult | 1

9. Primary Outcome: Number of Surgeon Responses to Optic Exchange Surgery Question: How Would You Rate the Surgical Difficulty of the Optic Implantation and Assembly (Exchange)? - Cohort 2
Description: as for outcome 7
Time Frame: Day 0 post-exchange
Population: as for outcome 7
Measure: Number; unit: surgeon response
Units Other Than Participants: eyes
Groups:
- Cohort 2: Subset of Cohort 1 with optic exchange at Month 1 post primary implantation, followed up to Month 1 post optic exchange
Arm/Group | Cohort 2
Number analyzed (Participants) | 4
Number analyzed (eyes) | 4
surgeon response
  Very easy | 1
  Easy | 1
  Neutral | 2

10. Primary Outcome: Number of Surgeon Responses to Optic Exchange Surgery Question: How Would You Rate the Surgical Difficulty of the Optic Disassembly? - Cohort 2
Description: as for outcome 7
Time Frame: Day 0 post-exchange
Population: as for outcome 7
Measure: Number; unit: surgeon response
Units Other Than Participants: eyes
Arm/Group | Cohort 2
Number analyzed (Participants) | 4
Number analyzed (eyes) | 4
surgeon response
  Very easy | 1
  Easy | 3

11. Primary Outcome: Number of Surgeon Responses to Optic Exchange Surgery Question: How Would You Rate the Surgical Difficulty of the Optic Explantation? - Cohort 2
Description: as for outcome 7
Time Frame: Day 0 post-exchange
Population: as for outcome 7
Measure: Number; unit: surgeon response
Units Other Than Participants: eyes
Arm/Group | Cohort 2
Number analyzed (Participants) | 4
Number analyzed (eyes) | 4
surgeon response
  Very easy | 1
  Easy | 1
  Neutral | 2

12. Primary Outcome: Number of Secondary Surgical Interventions (SSI) (Other Than Optic Exchange)
Description: A secondary surgical intervention (SSI) was defined as a surgical procedure that occurred after primary implantation and was conducted for the purpose of resolving residual refractive error (RRE) and optimizing visual outcomes, as determined by the investigator. No formal statistical hypothesis testing was planned.
Time Frame: Cohort 1: Up to one month post primary implantation, with one site followed up to 12 months. Cohort 2: Up to one month post exchange, for a total of up to 2 months.
Population: as for outcome 7
Measure: Number; unit: SSI
Units Other Than Participants: eyes
Arm/Group | All HMIOL Cohort
Number analyzed (Participants) | 78
Number analyzed (eyes) | 100
SSI | 4

13. Primary Outcome: Number of Device Deficiencies
Description: A device deficiency was defined as a failure of the device to meet its performance specifications or expectations, or otherwise not perform as intended. This could include either a malfunction or damage to the device or any part thereof, regardless of the source of malfunction or damage, including user error, and regardless of the presence of injury (or lack thereof) to subject, user, or bystander. No formal statistical hypothesis testing was planned.
Time Frame: as for outcome 12
Population: as for outcome 7
Measure: Number; unit: device deficiencies
Units Other Than Participants: eyes
Arm/Group | All HMIOL Cohort
Number analyzed (Participants) | 78
Number analyzed (eyes) | 100
device deficiencies | 4

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from time of consent to study exit: Cohort 1: Up to one month post primary implantation, with one site followed up to 12 months. Cohort 2: Up to one month post exchange, for a total of up to 2 months.
Description: AEs were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes.
Groups:
- Non-Ocular: All subjects with attempted HMIOL implantation (successful or aborted after contact with the eye)
- Ocular: All eyes with attempted HMIOL implantation (successful or aborted after contact with the eye)
Arm/Group | Non-Ocular | Ocular
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/100
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/100
Other Adverse Events (participants affected / at risk) | 0/78 | 12/100
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Non-Ocular (N=78) | Ocular (N=100)
Iridocyclitis (Eye disorders) | 0 | 6
Intraocular pressure increased (Investigations) | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT03681886/SAP_000.pdf
  • Study Protocol (2016-01-07): https://cdn.clinicaltrials.gov/large-docs/86/NCT03681886/Prot_001.pdf